CLINICAL TRIAL: NCT03100175
Title: Strength and Aerobic Training in Elderly Lymphoma Patients During Chemotherapy and Its Impact on Treatment Outcomes, Patients Functioning and Biological Markers of Ageing
Brief Title: Strength and Aerobic Training in Elderly Lymphoma Patients During Chemotherapy and Its Impact on Treatment Outcomes, Patients Functioning and Biological Markers of Aging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, IULIANA VAXMAN, principal investigator, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 113-17
Record Dates: First submitted 2017-03-06; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Strength Aerobic Training Elderly Lymphoma Sarcopenia Aging
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): the patient will be scheduled for another appointment and taught a set of exercises including strength training for upper and lower limbs (with elastic bands and weights, rising up from chair and climbing stairs), fitness work out (brisk walking) and balance exercises, as recommended by senior sport programs.
  * Patients will be provided with printed instructions explaining the recommended exercises, and with a diary to fill in, with days and number of repetitions of specific training elements to be checked in according to their compliance. Patients will also be equipped with a pedometer and will be asked to record the counts regularly
  * Patients will be met again by a physiotherapist for follow up at the start of every chemotherapy course (once in 3-4 weeks) and will be contacted by phone twice weekly to assure they stick to the training recommendations
  Interventions: Behavioral: physiotherapy
- control (No Intervention): The control group will receive standard treatment and follow-up with no special emphasis on physical activity

INTERVENTIONS:
Behavioral: physiotherapy — strength training for upper and lower limbs fitness and balance work out
  Arms: intervention

SUMMARY:
Frailty, one of geriatric syndromes, is considered a major obstacle for recovery from physiological stress. Such stress is imposed on patients with cancer by virtue of the disease itself but even more so by the treatment. Moreover, malignancy and chemotherapy both cause accelerated loss of muscle mass, deconditioning, frailty and negative outcomes. Several studies showed that chemotherapy accelerates ageing.

Muscle mass reserve was found to be a major predictor of outcomes in patients treated with chemotherapy. Recently, several studies suggest that active muscle strength training during chemotherapy may decrease side effects, improves the ability to deliver intended doses of treatment and may even affect oncological outcomes.

In the proposed study we intend to assess the contribution of physical training to the well-being of chemotherapy treated older patients, assessed by molecular and physiological parameters.

We intend to recruit lymphoma patients above age of 70 and prospectively and randomly assign them to the intervention group (strength, aerobic and balance training during the chemotherapy) and control group (standard care with no special emphasis on physical activity during the treatment).

We will measure clinical outcomes such as treatment tolerance and effects as well as physiological outcomes (muscle strength and mass, elements activities of daily living) and laboratory markers of ageing such as DNA methylation, INK 4a expression, telomere length and serum levels of inteleukin 6, CRP among others.

Our hypothesis is that physical training will improve patients' ability to complete the treatment with fewer side effects, will provide them with better daily functioning and better muscle strength/function. We also hypothesize that the ageing process, as shown by laboratory senescence markers, will be attenuated in the intervention group.

DETAILED DESCRIPTION:
Introduction Rising life expectancy and an exponential correlation between age and cancer incidence brought about a new field of geriatric oncology. As patients above age 65 account for more than 60% of cancer diagnoses with octogenarians and even nonagenarians being not rare in oncology practice, a geriatric prospective becomes essential in the treatment process.

Frailty, a nebulous term, defined on the metabolic basis as "vicious circle of energetic dysregulation", is largely heterogeneous in younger elderly population, with some people being frail, others borderline -"prefrail" or even non-frail - "fit". Nevertheless, frailty becomes universal as senescence progresses, as it is tightly linked with physiological ageing and usually worsened by comorbidities. Elderly patients can seem fit and in good health but still be "sub-clinically" frail. The clinical significance is a gradual loss of ability to cope and recover from physiological stress.

Oncological patients are exposed to two major physiological stresses: the catabolic state induced by the disease and the chemotherapy challenge to tissues.

Curative-intent chemotherapy is usually withheld from very frail individuals but elderly patients deemed to be pre-frail or fit are frequently treated according to standard or mildly modified protocols, putting them at risk of slow or no recovery from drug related toxicity. Moreover, it was shown in other studies that chemotherapy itself accelerates senescence by stress related mechanisms and promotes muscle loss and frailty in younger individuals .

Numerous tools have been developed to try to measure frailty and help treatment decisions. Despite some differences, the main bulk of evaluated elements in all of those tools refer in some way to patient's ability to perform physical activity including muscle strength, walking speed, level of energy production and feeling tired, emphasizing the critical role of muscles in elderly general condition .

Interventions shown to prevent deterioration and even improve physical condition of frail individuals were muscle training and nutritional support.

On the other hand, incorporation of physical training in younger oncological patients was shown to improve outcomes such as ability to complete chemotherapy without dose adjustment, subjective feeling of less fatigue, better daily functioning, earlier return to work and better physical measures of muscle strength and cardio-pulmonary fitness.

The positive impact of physical activity on both: preventing of frailty deterioration and ability to withstand chemotherapy better, led us to hypothesis that it would be especially beneficial in elderly cancer patients. The benefit would probably expand beyond the clinical and functional measures and would be also expressed on the molecular level with reduced levels of senescence markers.

We intend to prospectively recruit lymphoma patients above age of 70, admitted to Davidoff Cancer Center outpatient clinic and being judged eligible for chemotherapy at 75% of more of full dose. The patients will be randomly assigned to an intervention or control group. All patients will undergo a similar evaluation at the beginning and after completion of chemotherapy.

Standard evaluation of all patients:

* anthropomorphic measures (hand grip by a hand-held dynamometer and quadriceps strength by a sitting tensiometer), and functional measures (gait speed by 6 minute-walk, sit-to-stand test, functional reach and timed get-up-and-go test) - performed by a physiotherapist at the day of recruitment and one to two months after chemotherapy completion
* muscle mass according to muscle mass index calculation from the cross section area of both psoas muscles at the level of L3 vertebra corrected to height; and body composition according to mean Housfield units of the psoas section area - done by the study physician, using CT scans at the begging and after the treatment
* functional, nutritional and cognitive function as performed routinely at the Senior Oncology Program at Davidoff Cancer Center - done at the beginning and after the treatment by a team member
* standard blood tests including hemoglobin, white blood cells, albumin, CRP to be drawn before and after the treatment
* markers of senescence to be measured after the treatment completion: DNA methylation at three selected loci, expression of p16INK4A , telomere length and plasma levels of IL-6 and CRP - markers of "inflamm-aging" - a process of chronic low-level inflammation universal in older individuals.
* After the standard part of the evaluation by a physiotherapist, the patient will be scheduled for another appointment and taught a set of exercises including strength training for upper and lower limbs (with elastic bands and weights, rising up from chair and climbing stairs), fitness work out (brisk walking) and balance exercises, as recommended by senior sport programs.
* Patients will be provided with printed instructions explaining the recommended exercises, and with a diary to fill in, with days and number of repetitions of specific training elements to be checked in according to their compliance. Patients will also be equipped with a pedometer and will be asked to record the counts regularly
* Patients will be met again by a physiotherapist for follow up at the start of every chemotherapy course (once in 3-4 weeks) and will be contacted by phone twice weekly to assure they stick to the training recommendations The control group will receive standard treatment and follow-up with no special emphasis on physical activity.

The size of each group will be about 50 patients. Innovation To the best of our knowledge, there are no prospective studies published on this kind of intervention in elderly cancer patients. Home-based physical training is a simple, low-cost modality, which, if proven effective, would appreciably improve patient-related outcomes and probably reduce short and long-term costs of patient care. There are no studies that explored differences in cellular senescence in elderly cancer patient undergoing physical training.

Study design This will be a prospective randomized study, with an intervention to which no blinding can be done. The cross-sectional comparisons between the groups and longitudinal changes will be searched.

Statistics The statistical analysis of the data will be performed by a statistician of Rabin Medical Center using SPSS software and according to accepted standards.

ELIGIBILITY:
Inclusion Criteria:

* 70 years old and older
* Newly diagnosed large B cell lymphoma, Hodgkin lymphoma or follicular lymphoma planned for at least 75% of full dose chemotherapy
* preserved cognition or mild dementia
* Ability to perform physical activity

Exclusion Criteria:

* no

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2019-03-15 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
treatment tolerance | 6 month
  treatment dose density
muscle strength and mass | 6 month
  evaluated by physiotherapists
elements activities of daily living | 6 month
  evaluated by physiotherapists
DNA methylation | 6 month
  blood tests
INK 4a expression | 6 month
  blood test
telomere length | 6 month
  blood tests
serum levels of inteleukin 6 | 6 month
  blood tests
CRP | 6 month
  blood tests

IPD SHARING:
Plan to Share IPD: No
no paln to share data, study will be done in our center only